CLINICAL TRIAL: NCT04188847
Title: Apatinib Combined With Cisplatin and Paclitaxel as First-line Chemotherapy for Recurrent or Persistent Advanced Cervical Cancer: A Single Arm, Single Center, Open, Phase II Trial
Brief Title: First-line Chemotherapy for Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REPACC-1
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Recurrent Cervical Carcinoma; Persistent Advanced Cervical Carcinoma; Chemotherapy; Vascular Endothelial Growth Factor 2 Inhibitor; Apatinib; Targeted Therapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Drug Therapy; apatinib

STUDY DESIGN:
Intervention Model Description: A combination of cisplatin, paclitaxel and apatinib would be given for all patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): The patients would accept the regimen of apatinib combined with cisplatin and paclitaxel
  Interventions: Drug: Chemotherapy plus apatinib

INTERVENTIONS:
Drug: Chemotherapy plus apatinib — A combination of cisplatin, paclitaxel and apatinib would be given for all patients:
  * Cisplatin: 50 mg/m2 body surface area, on the first day, every 3 weeks. If the creatinine clearance rate was less than 40 ml/min, the cisplatin would be replace by carboplatin (area under ther curve = 5)
  * Paclitaxel: 50 mg/m2 body surface area, on the first day, every 3 weeks
  * Apatinib: 250 mg every day The total courses of cisplatin and paclitaxel would be no more than 6.
  Other Names: First line chemotherapy plus apatinib

SUMMARY:
The response rate of traditional first-line chemotherapy for recurrent or persistent advanced cervical cancer was low. This single arm, open, phase II trial would recruit 37 eligible patients. A combination of cisplatin, paclitaxel and apatinib would be given for first 23 patients. If at least 13 patients achieved complete or partial remission, the same regimen would be given for rest patients. The primary end is overall response rate (ORR). The second ends include progression-free survival, overall survival, disease control rate, remission duration, and adverse events. A molecular testing, mainly consisting of genomic analysis, will be carried in the oncologic tissues.

ELIGIBILITY:
Inclusion Criteria:

* Female of 18-75 years old
* Eastern Cooperative Oncology Group score 0-1
* Pathological confirmed of uterine cervical adenocarcinoma, squamous carcinoma, or adenosquamous carcinoma, with stage IA1 (with lymph-vascular space invasion) to IVB, which had accepted radical treatment for the purpose of cure
* An interval of 3 months or more since the fulfilling of last treatment
* At least one measurable lesion defined by Response Evaluation Criteria in Solid Tumors (RECIST) guideline 1.1
* Anticipative survival period of 3 months or more
* Lab testing within reference ranges
* With appropriate contraception
* Provided consents of participating the trial

Exclusion Criteria:

* With a history of exposure to other antiangiogenic agents
* With other malignancies within past 3 years
* With vital complications
* With uncontrolled hypertension despite of medical treatment
* With severe cardiac disease, coagulation disorders, bleeding disorders, vascular diseases, deep venous thrombosis
* With brain metastasis
* With addiction to psychiatric medications or with mental disorders
* With severe open trauma, fracture or major surgery with past 4 weeks
* With disorders which would hamper the absorption of oral drugs, or with intestinal perforation or ileus with past 6 months
* Urine protein ≥++, or 24 hr urine protein ≥1.0 g
* With potential allergy or intolerance to study regimens
* Not eligible for the study judged by researchers

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2022-02-06 (Actual); Study Completion 2022-03-13 (Actual)

PRIMARY OUTCOMES:
Overall response rate | One year
  The rates of complete and partial remission

SECONDARY OUTCOMES:
Progression-free survival | One year
  The length of time during and after the treatment of the cancer, that a patient lives with the disease but it does not get worse
Overall survival | One year
  The length of time from either the date of diagnosis or the start of treatment for the cancer, that patients diagnosed with the disease are still alive.
Disease control rate | One year
  The rates of complete and partial remission, and stable disease
Adverse event rates | One years
  The rates of adverse events judged by Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be available by public reports.
Supporting Information: Study Protocol, CSR
Time Frame: Two year
Access Criteria: Public reports